CLINICAL TRIAL: NCT02329886
Title: The Qingdao Port Health Study
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 20141218
Record Dates: First submitted 2014-12-20; First posted 2015-01-01 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Disease
Keywords: chronic diseases; risk factors; health outcomes
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In 2013, whole blood samples were collected for future genetic studies. And saliva and urine samples were also collected for future analysis.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
China, efforts are underway to respond to an unprecedented epidemiologic transition, with soaring rates of cardiovascular disease (CVD), including heart disease and stroke. Yet there may be limitations in translating observations and findings derived from Anglo-based population studies. As such, there is a critical need for population-based studies that provide insight into the risk factors, incidence, and outcomes of CVD in China. The Qingdao Port Health Study is a population-based prospective cohort study of employees of the Qingdao Port Group, China, designed to investigate the burden of CVD and risk factors (e.g., sociodemographic, biological, environmental and clinical factors) associated with disease onset and outcomes.

DETAILED DESCRIPTION:
In Qingdao Port, annual health assessments are offered at 3 on-site health clinics. The annual health assessment consists of a questionnaire, physical examination, laboratory tests, bio-sampling, and imaging examinations.In each year, demographics information, medical history, medication use and adherence, family history,lifestyles (e.g., nutritional intake; physical activity; smoking; alcohol use/abuse), menopause (including hormone use) and quality of life were collected by trained researchers.In 2013, blood and saliva samples were collected. Follow-up health assessments are performed every year. The outcomes of cardiovascular disease (angina, myocardial infarction, heart failure, stroke, revascularization), non-communicable diseases (chronic obstructive pulmonary disease, renal failure, liver disease and cancer), and all-cause death are collected from local medical insurance database.This study aim to surveillance of cardiovascular and other non-communicable diseases (risk factors, health outcomes and trends) and investigate of socio-cultural, biological, behavioral, social, and environmental factors on work performance, cardiovascular disease onset and cardiovascular health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All employees and retirees in Qingdao Port Group
* Aged over 18 years old

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Employees and retirees in Qingdao Port Group, Shandong province, China
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Actual)
Dates: Start 2013-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 3 year
  The number of all cause death will be collected. The effects of modified risk factors on all cause mortality will be assessed.

SECONDARY OUTCOMES:
Heart diseases (defined as myocardial infarction, agina requiring hospitalization and acute/chronic heart failure) | 3 year
  The number of heart disease outcomes will be collected because one person may have more than one time heart diseases. The incidence of heart disease is calculated by dividing the number of heart disease outcomes by the total number of participants in baseline study.
stroke (defined as ischemic stroke and hemorraghic stroke) | 3 year
  The number of stroke outcomes will be collected. The incidence of stroke is calculated by dividing the number of stroke outcomes by the total number of participants in baseline study.
revascularization (defined as percutaneous coronary intervention, coronary artery bypass grafting and percutaneous transluminal coronary angioplasty) | 3 year
  The number of revascularizations will be collected, one person may receive more than one time revascularizations. The incidence of revascularization is calculated by dividing the number of revascularization outcomes by the total number of participants in baseline study.

OTHER OUTCOMES:
chronic obstructive pulmonary disease | 3 year
  The number of participants with chronic obstructive pulmonary disease (COPD) will be collected. The incidence of COPD is calculated by dividing the number of COPD by the total number of participants in baseline study.
chronic renal insufficiency | 3 year
  The number of participants with chronic renal insufficiency will be collected. The incidence of chronic renal insufficiency is calculated by dividing the number of chronic renal insufficiency by the total number of participants in baseline study.
chronic liver diseases (defined as cirrhosis and hepatic failure) | 3 year
  The number of chronic liver diseases will be collected. The incidence of chronic liver diseases is calculated by dividing the number of chronic liver diseases by the total number of participants in baseline study.
cancer (defined as cancer, recurrence of cancer and cancer metastasis) | 3 year
  The number of cancer outcomes will be collected. The incidence of cancer is calculated by dividing the number of cancer outcomes by the total number of participants in baseline study.

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Jiang, MD, PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital; Xiancheng Liu, MD, PhD, Principal Investigator — Qingdao Fuwai hospital

REFERENCES:
- [Derived] Spatz ES, Jiang X, Lu J, Masoudi FA, Spertus JA, Wang Y, Li X, Downing NS, Nasir K, Du X, Li J, Krumholz HM, Liu X, Jiang L. Qingdao Port Cardiovascular Health Study: a prospective cohort study. BMJ Open. 2015 Dec 9;5(12):e008403. doi: 10.1136/bmjopen-2015-008403. PMID 26656011